CLINICAL TRIAL: NCT03391141
Title: In Vivo Aerodynamic Modeling of the Upper Airway in OSA
Brief Title: Diagnostic Validation of Drug-Induced Sleep Endoscopy (DISE)
Status: Completed | Type: Observational
Sponsor: Dr. Erica Thaler (Other)
Responsible Party: Sponsor-Investigator, Dr. Erica Thaler, Professor, University of Pennsylvania
Organization: University of Pennsylvania (Other)
Other Study IDs: 827621
Record Dates: First submitted 2017-12-08; First posted 2018-01-05 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Obstructive Sleep Apnea
Keywords: obstructive sleep apnea; sleep endoscopy; drug induced sleep endoscopy; diagnostic validation
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study aims to validate whether the pattern of airway collapse recorded during Drug-Induced Sleep Endoscopy (DISE) mirrors that of natural sleep, and to develop a model for airway collapse. Sensors will be placed in subjects' upper airways during DISE and then during in-lab sleep studies. The sleep study results will be compared with OR findings to create an aerodynamic model for natural sleep and to assess whether airway observations during DISE were valid representations of natural sleep.

DETAILED DESCRIPTION:
Drug-induced sleep endoscopy (DISE) was developed in 1991 as a technique to characterize upper airway collapse in patients with OSA. With the advent of various upper airway surgeries introduced in recent years, DISE has become increasingly utilized by the sleep surgeon as a surrogate for airway collapse during natural sleep in order to tailor a surgical approach for each patient. Propofol and/or midazolam infusions are typically used for sedation in these cases, however, there is limited evidence to suggest that these anesthetics reproduce natural sleep architecture. Therefore, it cannot be assumed that the pattern of collapse observed during DISE is reflective of natural sleep.

The aim of this study is to validate whether the pattern of collapse recorded during DISE mirrors that of natural sleep. Furthermore, the investigators aim to develop a quantitative in vivo model for airway collapse in order to further our understanding of the pathophysiology of OSA. They will do this by comparing the findings from DISE with aerodynamic readings from within the upper airway during natural sleep. The proposed technique will employ technologies already approved by the FDA for clinical use. Capacitance circuitry, airflow sensors, and/or pressure transducers will be suspended within the upper aerodigestive tract along a thin, low-profile, and flexible tube. During Phase I of the study, this aerodynamic probe will be placed in the OR during DISE along the upper airway, namely in the retropalatal, retroglossal, and hypopharyngeal regions. Readings will be correlated and calibrated with DISE findings in real-time. During Phase II, these sensors will again be placed within the same patients during in-office sleep studies. The results from the sleep study will be analyzed in conjunction with OR findings in order to create an aerodynamic model for natural sleep. This will also allow the investigators to assess whether airway observations during DISE were valid representations of natural sleep.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate to severe OSAS
* Must have symptoms of OSAS
* Must have sleep study showing AHI of 15 or greater
* Failed trial of CPAP
* BMI less than 35
* Be a surgical candidate for ablative or neuro-stimulation surgery
* Acceptable surgical comorbidities
* Non-aberrant upper airway anatomy
* Must demonstrate reliability in keep appointments

Exclusion Criteria:

* Prior ablative airway surgeries
* Allergies to oxymetazoline or lidocaine
* Significant central sleep apnea
* Presence of other sleep disorders
* History of neurologic or neuromuscular disease
* Historical or present substance abuse
* Bleeding disorders
* Autoimmune diseases that increase risk of nasal trauma such as Wegener's, Sarcoidosis, etc.
* Pregnancy
* Unacceptable anesthesia risk
* Ablative or orthognathic airway surgery
* Significant weight loss or weight gain with or without bariatric surgery
* Initiation of new drug that is known to alter sleep architecture
* Development of head and neck neoplasm
* Development of autoimmune disease altering airway anatomy
* Trauma to head and neck region

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with moderate to severe obstructive sleep apnea who have failed a trial of CPAP.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
site of airway obstruction | 3 months
  the presence or absence of airway obstruction in the retropalatal, retroglossal, and hypopharyngeal areas

CONTACTS AND LOCATIONS:
Overall Officials: Erica Thaler, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States